CLINICAL TRIAL: NCT01858948
Title: Risk and Protective Factors for SGA-induced Metabolic Syndrome in Bipolar Youth
Brief Title: SGA-induced Metabolic Syndrome in Bipolar Youth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robert McNamara, Associate Professor of Psychiatry, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK097599-01A1; 5R01DK097599 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Bipolar Youth Treated With Second-generation Antipsychotics
Keywords: Bipolar disorder; Second-generation antipsychotics; Obesity; Cardiometabolic risk
MeSH Terms: conditions — Bipolar Disorder; Obesity | interventions — Corn Oil; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine plus Omega (Experimental): Patients will be randomized to EPA+DHA supplements (OmegaRx) at fixed dose of 3.0 g/day (EPA: 2.0 g, DHA: 1.0 g; 5 capsules/d) for 24 weeks.
  Interventions: Drug: Omega; Drug: Quetiapine fumarate
- Quetiapine plus Placebo (Placebo Comparator): Patients will be randomized to similar in shape an color placebo supplements (corn oil)
  Interventions: Drug: Placebo; Drug: Quetiapine fumarate

INTERVENTIONS:
Drug: Omega — Omega-3 supplements
  Other Names: EPA+DHA supplements (OmegaRx)
  Arms: Quetiapine plus Omega
Drug: Placebo — Similar in shape and color to Omega supplements
  Other Names: Placebo supplements (corn oil) provided by the Inflammation Research Foundation
  Arms: Quetiapine plus Placebo
Drug: Quetiapine fumarate — Prior to randomization to Omega/placebo, patients were started on 100 mg BID of quetiapine, and the dose adjusted based on tolerability and response. The quetiapine target dose is 400-600 mg.
  Other Names: Seroquel

SUMMARY:
The investigators tested the hypothesis that long-chain omega-3 (LCn-3) fatty acid supplementation will attenuate the adverse cardiometabolic effects of second-generation antipsychotics exposure in first-episode adolescent manic patients.

DETAILED DESCRIPTION:
Following acute (6-week) open-label treatment with quetiapine, first-episode adolescent manic patients (ages 10-17 years) were randomized to double-blind adjunctive treatment with long-chain omega-3 (LCn-3) fatty acids or placebo for 24 weeks to investigate protective effects on the of adverse cardiometabolic events and weight gain during quetiapine maintenance therapy. They will have 6 visits over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR criteria for bipolar disorder, type I, manic or mixed episode
* Baseline YMRS score > 20
* Ages 10-17 years
* Tanner scale stages III-V
* No prior exposure to SGA medications
* Fluent in English
* Provision of written informed consent by a legal guardian and written assent by the subject
* Manic or depressive symptoms do not result entirely from acute medical illness or acute intoxication or withdrawal from drugs or alcohol as determined by medical evaluation and rapid symptom resolution
* If female and of child bearing potential, agrees to use one of the following method of birth control: complete abstinence from sexual intercourse, barrier (diaphragm or condom), or oral/injectable contraceptive. For Phase II, additional Inclusion criteria are
* Receiving a stable therapeutic dose of quetiapine for a minimum of 1 week (i.e., patients who achieved remission (YMRS total score 7 during Phase I)
* Not requiring concomitant use of antidepressant or mood-stabilizer medications (see Section C.4.c. Concomitant Medications).

Exclusion Criteria:

* IQ < 70, as determined by The Wechsler Abbreviated Scale of Intelligence
* Positive pregnancy test (to avoid teratogenesis)
* A history of major cardiovascular or neurological illness
* Any lifetime DSM-IV-TR substance use disorder (nicotine dependence is permitted)
* A lifetime DSM-IV-TR diagnosis of any pervasive developmental disorder
* Any history of a hematological disorder in themselves or a first-degree relative will be excluded (since omega-3 fatty acids may be associated with anti-thrombotic effects). Similarly, concomitant use of medications with anticoagulant effects (e.g. aspirin) will be prohibited
* Allergy to fish/seafood; 8) Currently taking omega-3 fatty acid supplements

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2013-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients received 6-week open-label quetiapine prior to entering the trial.
Groups:
- Quitiapine Plus Omega: Patients will be randomized to EPA+DHA supplements (OmegaRx) at a fixed dose of 3.0 g/day (EPA: 2.0 g, DHA: 1.0 g; 5 capsules/d) for 24 weeks
  Omega: Omega-3 supplements
  Quetiapine fumarate: Patients will be started on 100 mg BID of quetiapine, and the dose adjusted based on tolerability and response. The quetiapine target dose is 400-600 mg.
- Quetiapine Plus Placebo: Patients will be randomized to similar in shape an color placebo supplements (corn oil)
  Placebo: Similar in shape and color to Omega supplements
  Quetiapine fumarate: Patients will be started on 100 mg BID of quetiapine, and the dose adjusted based on tolerability and response. The quetiapine target dose is 400-600 mg.
Period: Overall Study
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo
Started | 9 | 10
Completed | 5 (Completed week 24) | 4 (Completed week 24)
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Quitiapine Plus Omega: Patients will be randomized to EPA+DHA supplements (OmegaRx) a fixed dose of 3.0 g/day (EPA: 2.0 g, DHA: 1.0 g; 5 capsules/d) for 24 weeks
  Omega: Omega-3 supplements
  Quetiapine fumarate: Patients will be started on 100 mg BID of quetiapine, and the dose adjusted based on tolerability and response. The quetiapine target dose is 400-600 mg.
- Total: Total of all reporting groups
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (2.2) | 14.1 (1.8) | 14.7 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (4.2) | 26.2 (6.1) | 24.7 (5.4)
Fasting blood triglyceride levels [Mean (Standard Deviation); unit: mg/dL] | 122.3 (43.5) | 122.9 (54.9) | 122.6 (47.1)
Manic Symptom Severity [Mean (Standard Deviation); unit: units on a scale] | 26.2 (6.6) | 21.1 (7.6) | 23.5 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI) is a measure of body fat calculated as weight in kilograms divided by height in meters squared (kg/m^2). BMI Categories are:
  Underweight = <18.5; Normal weight = 18.5-24.9; Overweight = 25-29.9; Obesity = BMI of 30 or greater. Greater decreases in BMI are a better outcome.
Time Frame: 24 weeks
Population: First-episode adolescent manic patients treated with open-label quetiapine were randomized to adjunctive treatment with fish oil or placebo for 24-weeks.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Quitiapine Plus Omega: Patients will be randomized to EPA+DHA supplements (OmegaRx) for 24 weeks
  Omega: Omega-3 supplements
  Quetiapine fumarate: Patients will be started on 100 mg BID of quetiapine, and the dose adjusted based on tolerability and response. The quetiapine target dose is 400-600 mg.
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo
Number analyzed (Participants) | 9 | 10
kg/m^2 | 24.4 (4.7) | 26.3 (7.4)

2. Primary Outcome: Fasting Blood Triglycerides Levels
Description: Triglycerides are the chemical form in which most fat exists in food as well as in the body. They're also present in blood plasma and, in association with cholesterol, form the plasma lipids. Levels are categorized as follows: Normal - Less than 150 milligrams per deciliter (mg/dL); Borderline high - 150 to 199 mg/dL; High - 200 to 499 mg/dL; Very high - 500 mg/dL or above. Greater reductions blood triglyceride levels are a better outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo
Number analyzed (Participants) | 9 | 10
mg/dL | 99.7 (24.9) | 88 (39.3)

3. Secondary Outcome: Manic Symptom Severity
Description: Manic symptom ratings will be obtained using the Young Mania Rating Scale (YMRS). The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania: Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania). Greater reductions from baseline indicates a greater improvement in manic symptoms.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo
Number analyzed (Participants) | 9 | 10
units on a scale | 4.3 (3.7) | 7.2 (5.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Quitiapine Plus Omega | Quetiapine Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT01858948/Prot_SAP_000.pdf